CLINICAL TRIAL: NCT05558436
Title: Comparison of Diagnostic Sensitivity Between Circulating Tumor DNA Methylation and Carcinoembryonic Antigen in Colorectal Cancer
Brief Title: Comparison of Diagnostic Sensitivity Between ctDNA Methylation and CEA in Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-245
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Tumor
Keywords: colorectal cancer; advanced adenoma; circulating tumor DNA methylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Fresh plasma and tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with colorectal cancer and advanced adenoma.
  Interventions: Diagnostic Test: Genome-wide methylation profiling
- Control group: Healthy participants and patients with benign colorectal disease.
  Interventions: Diagnostic Test: Genome-wide methylation profiling

INTERVENTIONS:
Diagnostic Test: Genome-wide methylation profiling — Detection for colorectal tumor-specific ctDNA methylation biomarkers

SUMMARY:
This is a prospective diagnostic study. This study is to compare the performance between circulating tumor DNA (ctDNA) methylation and carcinoembryonic antigen (CEA) in detecting colorectal tumor. Firstly, based on the identification of differential ctDNA methylation biomarkers, the diagnostic model is established and the diagnostic performance was compared with that of CEA. Secondly, the stage stratification model was established preliminarily based on differential ctDNA methylation biomarkers and the performance was also compared with that of CEA.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide, the second deadliest cancer. It is reported that patients prefer non-invasive methods rather than invasive methods for the detection of CRC. Carcinoembryonic antigen (CEA) is commonly employed in clinical practice for early detection of CRC, but it is limited for its low sensitivity, which is around 30%-40%. DNA methylation is a commonly used biomarker for non-invasive tumor detection in plasma. We aim to develop and validate a ctDNA methylation-based blood test for CRC diagnosis based on genome-wide methylation detection. There are two steps in the study. Firstly, this prospective study aims to identify colorectal tumor differential circulating tumor DNA (ctDNA) methylation biomarkers, establish the diagnostic model. Secondly, we performed a preliminary study to stratify early-stage and advanced-stage disease based on the differential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Case group

* Patients must have histologically confirmed colorectal cancer or advanced adenoma.
* Patients need to receive surgical resection or endoscopic resection.
* Patients have a performance status of ≤1 on the ECOG Performance Scale.
* Written informed consent must be obtained.

Control group

* Written informed consent must be obtained.
* Individuals must receive colonoscopy.

Exclusion Criteria:

* Patients received tumor treatment prior to the drawn of blood sample, including surgical resection, neoadjuvant chemoradiotherapy and targeted therapy.
* Patients received antibiotics regularly.
* Patients received blood transfusion two weeks before the drawn of blood sample.
* Patients with indications of emergency surgery, including bleeding, obstruction and perforation.
* Patients who are positive for Human Immunodeficiency Virus (HIV).
* Patients with abnormal liver and kidney function.
* Patients with the history of other malignancies, inflammatory bowel disease and Lynch syndrome.
* Patients who are pregnant or breastfeeding.
* Alcoholic or drug abusers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | 3 years
  The comparison of sensitivity between ctDNA methylation and CEA in detecting colorectal cancer

SECONDARY OUTCOMES:
Stage stratification | 3 years
  The performance of the novel model to stratify early-stage and advanced-stage disease, and comparing with that of CEA.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D., Ph.D., Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Schilsky RL, Nass S, Le Beau MM, Benz EJ Jr. Progress in Cancer Research, Prevention, and Care. N Engl J Med. 2020 Sep 3;383(10):897-900. doi: 10.1056/NEJMp2007839. No abstract available. PMID 32877579
- [Background] Adler A, Geiger S, Keil A, Bias H, Schatz P, deVos T, Dhein J, Zimmermann M, Tauber R, Wiedenmann B. Improving compliance to colorectal cancer screening using blood and stool based tests in patients refusing screening colonoscopy in Germany. BMC Gastroenterol. 2014 Oct 17;14:183. doi: 10.1186/1471-230X-14-183. PMID 25326034
- [Background] Luo H, Zhao Q, Wei W, Zheng L, Yi S, Li G, Wang W, Sheng H, Pu H, Mo H, Zuo Z, Liu Z, Li C, Xie C, Zeng Z, Li W, Hao X, Liu Y, Cao S, Liu W, Gibson S, Zhang K, Xu G, Xu RH. Circulating tumor DNA methylation profiles enable early diagnosis, prognosis prediction, and screening for colorectal cancer. Sci Transl Med. 2020 Jan 1;12(524):eaax7533. doi: 10.1126/scitranslmed.aax7533. PMID 31894106
- [Background] Grotowski M. [Antigens (CEA and CA 19-9) in diagnosis and prognosis colorectal cancer]. Pol Merkur Lekarski. 2002 Jan;12(67):77-80. Polish. PMID 11957811
- [Background] Kanwal R, Gupta K, Gupta S. Cancer epigenetics: an introduction. Methods Mol Biol. 2015;1238:3-25. doi: 10.1007/978-1-4939-1804-1_1. PMID 25421652
- [Background] Shen SY, Singhania R, Fehringer G, Chakravarthy A, Roehrl MHA, Chadwick D, Zuzarte PC, Borgida A, Wang TT, Li T, Kis O, Zhao Z, Spreafico A, Medina TDS, Wang Y, Roulois D, Ettayebi I, Chen Z, Chow S, Murphy T, Arruda A, O'Kane GM, Liu J, Mansour M, McPherson JD, O'Brien C, Leighl N, Bedard PL, Fleshner N, Liu G, Minden MD, Gallinger S, Goldenberg A, Pugh TJ, Hoffman MM, Bratman SV, Hung RJ, De Carvalho DD. Sensitive tumour detection and classification using plasma cell-free DNA methylomes. Nature. 2018 Nov;563(7732):579-583. doi: 10.1038/s41586-018-0703-0. Epub 2018 Nov 14. PMID 30429608
- [Background] Xu RH, Wei W, Krawczyk M, Wang W, Luo H, Flagg K, Yi S, Shi W, Quan Q, Li K, Zheng L, Zhang H, Caughey BA, Zhao Q, Hou J, Zhang R, Xu Y, Cai H, Li G, Hou R, Zhong Z, Lin D, Fu X, Zhu J, Duan Y, Yu M, Ying B, Zhang W, Wang J, Zhang E, Zhang C, Li O, Guo R, Carter H, Zhu JK, Hao X, Zhang K. Circulating tumour DNA methylation markers for diagnosis and prognosis of hepatocellular carcinoma. Nat Mater. 2017 Nov;16(11):1155-1161. doi: 10.1038/nmat4997. Epub 2017 Oct 9. PMID 29035356
- [Background] Xie H, Mahoney DW, Foote PH, Burger KN, Doering KA, Taylor WR, Then SS, Cao X, McGlinch M, Berger CK, Wu TT, Hubbard JM, Allawi HT, Kaiser MW, Lidgard GP, Ahlquist DA, Kisiel JB. Novel Methylated DNA Markers in the Surveillance of Colorectal Cancer Recurrence. Clin Cancer Res. 2021 Jan 1;27(1):141-149. doi: 10.1158/1078-0432.CCR-20-2589. Epub 2020 Oct 7. PMID 33028593
- [Background] Cai G, Cai M, Feng Z, Liu R, Liang L, Zhou P; ColonAiQ Group; Zhu B, Mo S, Wang H, Lan X, Cai S, Xu Y, Wang R, Dai W, Han L, Xiang W, Wang B, Guo W, Zhang L, Zhou C, Luo B, Li Y, Nie Y, Ma C, Su Z. A Multilocus Blood-Based Assay Targeting Circulating Tumor DNA Methylation Enables Early Detection and Early Relapse Prediction of Colorectal Cancer. Gastroenterology. 2021 Dec;161(6):2053-2056.e2. doi: 10.1053/j.gastro.2021.08.054. Epub 2021 Sep 4. No abstract available. PMID 34487783
- [Background] Liang N, Li B, Jia Z, Wang C, Wu P, Zheng T, Wang Y, Qiu F, Wu Y, Su J, Xu J, Xu F, Chu H, Fang S, Yang X, Wu C, Cao Z, Cao L, Bing Z, Liu H, Li L, Huang C, Qin Y, Cui Y, Han-Zhang H, Xiang J, Liu H, Guo X, Li S, Zhao H, Zhang Z. Ultrasensitive detection of circulating tumour DNA via deep methylation sequencing aided by machine learning. Nat Biomed Eng. 2021 Jun;5(6):586-599. doi: 10.1038/s41551-021-00746-5. Epub 2021 Jun 15. PMID 34131323
- [Derived] Ji H, Xu M, Hu Y, Yan B, Wu W, Zheng J, Yan J. Preoperative Identification of Lymph Node Metastasis in Colorectal Cancer Using Noninvasive ctDNA Methylation Signatures: Results from a Prospective Study. Dis Colon Rectum. 2025 Dec 11. doi: 10.1097/DCR.0000000000004089. Online ahead of print. PMID 41378988